CLINICAL TRIAL: NCT01581281
Title: Amitriptyline and Topiramate in the Prevention of Childhood Migraine
Brief Title: The Childhood and Adolescent Migraine Prevention Study
Acronym: CHAMP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim assessment provided sufficient data to answer study questions
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIN-001; 1U01NS076788-01 (NIH)
Record Dates: First submitted 2011-12-16; First posted 2012-04-20 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-07

CONDITIONS: Migraine; Migraine Disorders; Headache
Keywords: Pediatric; Children; Adolescent; Headache; Migraine
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Amitriptyline; Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Amitriptyline (Active Comparator): Drug to be administered twice daily.
  Interventions: Drug: Amitriptyline
- Topiramate (Active Comparator): Drug to be administered twice daily.
  Interventions: Drug: Topiramate
- Placebo (Placebo Comparator): To be administered twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amitriptyline — Amitriptyline will be administered twice daily at home during the 8-week titration period followed by a 16 week maintenance phase of the highest tolerated dose. The morning dose is a placebo pill. Dosing of amitriptyline will be weight-based.
  Arms: Amitriptyline
Drug: Topiramate — Topiramate will be administered twice daily at home during the 8-week titration period followed by a 16 week maintenance phase of the highest tolerated dose. Dosing of topiramate will be weight-based.
  Arms: Topiramate
Drug: Placebo — Placebo will be administered twice daily at home during the 8-week titration period followed by a 16 week maintenance period.
  Arms: Placebo

SUMMARY:
The purpose of this research study is to test two medicines for migraine prevention in children and adolescents.

DETAILED DESCRIPTION:
The purpose of this research study is to test two medicines for migraine prevention in children and adolescents. The investigators want to see if amitriptyline and/or topiramate are better than placebo (sugar pill) in reducing headache frequency in children and adolescents ages 8 to 17 with migraines. At this time, there are no FDA approved medicines approved in the US for the prevention treatment of migraine headaches in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Migraine with or without aura (International Classification of Headache Disorders, 2nd Edition (ICHD-II) or chronic migraine (ICHD-II revised)
* Migraine frequency based upon prospective headache diary of 28 days must be ≥ 4. Migraine frequency defined as any migraine during one day in the 28 day baseline period (1)
* PedMIDAS Disability Score > 10, indicating at least mild disruption in daily activities and < 140, indicating extreme disability that may require more comprehensive, multi-component therapy
* Females or males 8-17 years, inclusive

  1. Migraine frequency is defined as the period from the onset to the stop time of painful migraine symptoms not to exceed 24 hours with the clock starting at midnight. If painful symptoms last longer than 24 hours, this is considered a new and distinct migraine headache. If painful symptoms recur within 24 hours of initial onset, this is considered part of the initial migraine episode and would be counted as one migraine.

Exclusion Criteria:

* Continuous migraine defined as an unrelenting headache for a 28 day period
* Weight less than 30 kg or greater than 120 kg
* Unwilling to avoid taking non-specific acute medication such as NSAIDS (e.g., ibuprofen), more than 3 times per week, or migraine specific acute medications such as triptans more than 6 times per month
* Currently taking other prophylactic anti-migraine medication within a period equivalent to 2 weeks of that medication before entering the screening phase, or the use of Botulinum toxin (Botox®) within 3 months of entering the screening phase
* Subjects who have previously failed an adequate trial of AMI or TPM for prophylaxis of at least 3 months duration at doses recommended for migraine relief because of lack of efficacy or adverse events(2)
* Current use of disallowed medications/products: opioids, antipsychotics, antimanics, barbiturates, benzodiazepines, muscle relaxants, sedatives, tramadol, nutraceuticals, SSRIs, or SSNRIs
* Known history of allergic reaction or anaphylaxis to AMI or TPM
* Abnormal findings on ECG at baseline, particularly lengthening of the QT interval greater than or equal to 450 msec
* Subject is pregnant or has a positive pregnancy test
* Subject is sexually active and not using a medically acceptable form of contraception
* Diagnosis of epilepsy or other neurological diseases
* History of kidney stones
* Inability to swallow pills after using behavioral techniques if indicated between screening visit and baseline visit (3)
* Present psychiatric disease as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM IV) (e.g. psychosis, bipolar disorder, major depression, generalized anxiety disorder), alcohol or drug dependence, or documented developmental delays or impairments (e.g., autism, cerebral palsy, or mental retardation) that, in the opinion of the site investigator, would interfere with adherence to study requirements or safe participation in the trial
* Any and all other diagnoses or conditions which in the opinion of the site investigator, that would prevent the patient from being a suitable candidate for the study or interfere with the medical care needs of the study subject

  (2)"Previously failed an adequate trial of AMI or TPM" is defined as: dosage of 1mg/kg/day of AMI or 2 mg/kg/day of TPM; trial of at least 3 months duration; efficacy of having at least a 50% decrease in migraine frequency in response to drug therapy; or unable to tolerate taking the medication due to treatment-related side effects.

  (3)Subjects who cannot swallow pills at the time of the screening visit will be given a training session using behavioral techniques. Upon return for baseline visit, if the subject continues to be unable to swallow pills, the subject will be excluded from the study.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 488 (Actual)
Dates: Start 2012-06; Primary Completion 2015-04 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott W. Powers, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Andrew D. Hershey, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Christopher S. Coffey, PhD, Principal Investigator — University of Iowa
Locations (35):
- United States (35):
  - Phoenix Children's Medical Group, Phoenix, Arizona
  - University of California-San Francisco Headache Center, San Francisco, California
  - Stanford Hospital and Clinics, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Premiere Research Institute, West Palm Beach, Florida
  - Atlanta Headache Specialists, Atlanta, Georgia
  - Josephson Wallack Munshower Neurology Research, Indianapolis, Indiana
  - Children's Mercy Hospital, Kansas City, Kansas
  - University of Louisville Health Sciences Center, Louisville, Kentucky
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Children's Hospital of Boston, Waltham, Massachusetts
  - New England Regional Headache Center, Worcester, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Saint Louis University, St Louis, Missouri
  - University of Nevada, Reno, Nevada
  - Dent Neurological Institute, Amherst, New York
  - Winthrop University Hospital, Mineola, New York
  - The Headache Institute at Roosevelt Hospital, New York, New York
  - Schenectady Neurological Constultants, PC, Schenectady, New York
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital, Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oklahoma Health Sciences, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Preferred Clinical Research, Pittsburgh, Pennsylvania
  - LeBonheur Children's Hospital, Memphis, Tennessee
  - Dallas Pediatric Neurology Associates, Dallas, Texas
  - Scott and White Healthcare, Temple, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Marshfield Clinic, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets and associated documentation will be submitted to NINDS for archiving and public access, consistent with current NINDS data sharing policy.

REFERENCES:
- [Derived] Reidy BL, Powers SW, Coffey CS, Chamberlin LA, Ecklund DJ, Klingner EA, Yankey JW, Korbee LL, Porter LL, Peugh J, Kabbouche MA, Kacperski J, Hershey AD; CHAMP Investigators. Multimodal Assessment of Medication Adherence Among Youth With Migraine: An Ancillary Study of the CHAMP Trial. J Pediatr Psychol. 2022 Apr 8;47(4):376-387. doi: 10.1093/jpepsy/jsab123. PMID 34865085
- [Derived] Reidy BL, Peugh J, Hershey AD, Coffey CS, Chamberlin LA, Ecklund DJ, Klingner EA, Yankey JW, Korbee LL, Porter LL, Kabbouche MA, Kacperski J, Powers SW. Trajectory of treatment response in the child and adolescent migraine prevention (CHAMP) study: A randomized clinical trial. Cephalalgia. 2022 Jan;42(1):44-52. doi: 10.1177/03331024211033551. Epub 2021 Aug 17. PMID 34404270
- [Derived] Powers SW, Coffey CS, Chamberlin LA, Ecklund DJ, Klingner EA, Yankey JW, Korbee LL, Porter LL, Hershey AD; CHAMP Investigators. Trial of Amitriptyline, Topiramate, and Placebo for Pediatric Migraine. N Engl J Med. 2017 Jan 12;376(2):115-124. doi: 10.1056/NEJMoa1610384. Epub 2016 Oct 27. PMID 27788026
- [Derived] Hershey AD, Powers SW, Coffey CS, Eklund DD, Chamberlin LA, Korbee LL; CHAMP Study Group. Childhood and Adolescent Migraine Prevention (CHAMP) study: a double-blinded, placebo-controlled, comparative effectiveness study of amitriptyline, topiramate, and placebo in the prevention of childhood and adolescent migraine. Headache. 2013 May;53(5):799-816. doi: 10.1111/head.12105. Epub 2013 Apr 17. PMID 23594025

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 16, 2012 through November 24, 2014, 488 patients were assessed for eligibility from 31 sites in the United States. Of those, 361 patients underwent randomization.
Pre-assignment Details: Of the patients assessed for eligibility, 21 (4%) did not undergo randomization owing to early trial closure and 106 (22%) were excluded. Eighty-one (81) were excluded due to not meeting inclusion criteria, 25 declined participation (13 were unwilling, but eligibility was otherwise confirmed and 12 were willing and eligibility was unknown).
Groups:
- Topiramate: Topiramate enclosed in capsules to maintain the blind was administered orally in a divided dose of 1 capsule twice daily. A target dose was 2 mg per kilogram per day. Dose escalation occurred every two weeks over a period of 8 weeks, with dose modification based on side effects. A 16 week constant-dose (maintenance) phase followed at the highest dosage achieved.
- Placebo: Placebo enclosed in capsules to maintain the blind was administered orally twice daily during an 8 week titration period followed by a 16 week maintenance phase (mirroring the other two treatment arms).
- Amitriptyline: Amitriptyline enclosed in capsules to maintain the blind was administered orally in dose of 1 capsule twice daily (AM capsule did not contain medication. A target dose was 1 mg per kilogram per day. Dose escalation occurred every two weeks over a period of 8 weeks, with dose modification based on side effects. A 16 week constant-dose (maintenance) phase followed at the highest dosage achieved.
Period: Overall Study
Arm/Group | Topiramate | Placebo | Amitriptyline
Started | 145 | 72 | 144
Completed | 130 | 66 | 132
Not Completed | 15 | 6 | 12
Not completed — Early Study Closure | 15 | 6 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topiramate | Placebo | Amitriptyline | Total
Number analyzed (Participants) | 145 | 72 | 144 | 361
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 145 | 72 | 144 | 361
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.2 (2.5) | 14.2 (2.2) | 14.2 (2.4) | 14.2 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 49 | 97 | 247
  Male | 44 | 23 | 47 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 6 | 8 | 28
  Not Hispanic or Latino | 123 | 65 | 128 | 316
  Unknown or Not Reported | 8 | 1 | 8 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 14 | 5 | 8 | 27
  Asian | 6 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 24 | 17 | 26 | 67
  White | 98 | 48 | 107 | 253
  More than one race | NA — data not collected | NA — data not collected | NA — data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 2 | 2 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 145 | 72 | 144 | 361
Headache Days [Mean (Standard Deviation); unit: days] — Number of headache days during 28-day baseline period
  days | 11.5 (6.1) | 11.0 (6.3) | 11.5 (6.2) | 11.4 (6.1)
Pediatric Migriane Disability Assessment Score (PedMIDAS) [Mean (Standard Deviation); unit: units on a scale] — Scores on the PedMIDAS range from 0 to 240, with a score of 1 to 10 indicating no disability, 11 to 30 indicating mild disability, 31 to 50 indicating moderate disability, and more than 50 indicating severe disability.
  units on a scale | 42.6 (27.4) | 42.9 (26.7) | 40.6 (26.4) | 41.9 (26.8)

OUTCOME MEASURES:

1. Primary Outcome: Number (Percentage) of Participants Reporting a ≥ 50% Reduction in Headache Days
Description: The primary endpoint was a ≥ 50% reduction in headache frequency from the 28 days (4 weeks) baseline period prior to randomization to the last 28 days (4 weeks) of the trial. Headache frequency was defined as the number of days with headache for a given four week 28 day (4 week) period. A headache day was defined as any day during which any headache occurs within a 24 hour period, starting and ending at midnight.
  For each participant, the primary endpoint involved a determination of whether a 50% or greater reduction in headache frequency was observed during the last 4 weeks of active treatment as compared with the headache frequency during the 4-week baseline period. Results were compared across the three treatment groups.
Time Frame: 4 week baseline period and last 4 weeks of the 24-week trial
Population: The primary endpoint involved a determination of whether a 50% or greater reduction in headache frequency was observed during the last 4 weeks of active treatment as compared with the headache frequency during the 4-week baseline period between the participants receiving amitriptyline and participants receiving placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Topiramate | Placebo | Amitriptyline
Number analyzed (Participants) | 130 | 66 | 132
Participants | 72 | 40 | 69
Statistical Analysis 1: Comparison: Placebo vs Amitriptyline; Logistic regression models were used to estimate the odds of successful primary endpoint for amitriptyline relative to placebo. The analyses followed the intention to treat principle, imputing an outcome of "failure" for any participant who withdrew early for any reason or did not provide week 24 headache diary data (endpoint data). The models, and corresponding odds ratios, were adjusted for the two stratification variables (age and baseline number of headache days); Test type: Superiority; p = 0.2636, Regression, Logistic — A Bonferroni approach was used to control the type I error rate. Because there were three comparisons, the Bonferroni corrected level of significance is 0.017 (= 0.05 / 3); Odds Ratio (OR) = 0.71, 98.3% CI 2-sided [0.34 to 1.48]
Statistical Analysis 2: Comparison: Topiramate vs Placebo; Logistic regression models were used to estimate the odds of successful primary endpoint for topiramate relative to placebo. The analyses followed the intention to treat principle, imputing an outcome of "failure" for any participant who withdrew early for any reason or did not provide week 24 headache diary data (endpoint data). The models, and corresponding odds ratios, were adjusted for the two stratification variables (age and baseline number of headache days); Test type: Superiority; p = 0.4821, Regression, Logistic — A Bonferroni approach was used to control the type I error rate. Because there were three comparisons of interest, the Bonferroni corrected level of significance is 0.017 ( = 0.05 / 3); Odds Ratio (OR) = 0.81, 98.3% CI 2-sided [0.39 to 1.68]
Statistical Analysis 3: Comparison: Topiramate vs Amitriptyline; Logistic regression models were used to estimate the odds of successful primary endpoint for topiramate relative to amitriptyline. The analyses followed the intention to treat principle, imputing an outcome of "failure" for any participant who withdrew early for any reason or did not provide week 24 headache diary data (endpoint data). The models, and corresponding odds ratios, were adjusted for the two stratification variables (age and baseline number of headache days); Test type: Superiority; p = 0.6107, Regression, Logistic — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 0.88, 98.3% CI 2-sided [0.49 to 1.59]

2. Secondary Outcome: Change in Absolute Headache Disability Score on PedMIDAS
Description: The PedMIDAS scale which evaluated the impact of headaches in school, home, play, and social activities, is comprised of six items that pertain to days missed in various activities over the past 90 days. Questions were answered by the youth in consultation with their parents and reviewed by study staff. The PedMIDAS scale was administered at baseline (covering the three months prior to enrollment) and at the 24-week endpoint visit (the end of the maintenance period, covering three months of enrollment). A total PedMIDAS score (sum of items 1-6) was used in this trial. Scores range from 0-240; with a score of 0-10 indicating no disability, 11-30 mild disability, 31-50 moderate disability, and more than 50 severe disability in daily activities. The main outcome measure for this comparison will be the difference in the baseline and endpoint (24 week) PedMIDAS total scores for:
  1. Amitriptyline vs. Placebo
  2. Topiramate vs. Placebo
  3. Amitriptyline vs Topiramate
Time Frame: baseline and 24 week endpoint
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Topiramate | Placebo | Amitriptyline
Number analyzed (Participants) | 130 | 66 | 132
units on a scale | -26.8 (27.5) | -22.6 (29.42) | -22.5 (26.37)
Statistical Analysis 1: Comparison: Placebo vs Amitriptyline; The mean change from baseline in PedMIDAS score over time for the three groups was assessed using a linear regression model for each of the three pairwise comparisons (Amitriptyline relative to placebo, Topiramate relative to placebo, and Amitriptyline relative to Topiramate), adjusted for the baseline PedMIDAS score. The models, and corresponding odds ratios, were adjusted for the two stratification variables (age and baseline number of headache days); Test type: Superiority; p = 0.9137, Regression, Linear; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-6.64 to 5.95]
Statistical Analysis 2: Comparison: Topiramate vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1331, Regression, Linear; Median Difference (Final Values) = -4.84, 95% CI 2-sided [-11.16 to 1.49]
Statistical Analysis 3: Comparison: Topiramate vs Amitriptyline; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1011, Regression, Linear; Mean Difference (Final Values) = 4.49, 95% CI 2-sided [-0.88 to 9.87]

3. Secondary Outcome: Change in Number of Headache Days
Description: This outcomes measure examines whether the rate of absolute number of headache days, per 28 day period, differs between treatment groups over time. This was assessed longitudinally based on the actual number of headache days from the 28 days prior to randomization to the last 28 days of this 24 week trial. The change in absolute headache days was compared between:
  1. Amitriptyline vs. placebo
  2. Topiramate vs. placebo
  3. Amitriptyline vs. Topiramate
Time Frame: 4 week baseline period and last 4 weeks of the 24-week trial
Population: The analysis population included all participants who had observed end-point data: 101 in the topiramate group, 59 in the placebo group, and104 in the amitriptyline group.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Topiramate | Placebo | Amitriptyline
Number analyzed (Participants) | 101 | 59 | 104
days | -6.7 (4.99) | -5.9 (6.96) | -6.7 (6.20)
Statistical Analysis 1: Comparison: Placebo vs Amitriptyline; Another major secondary objective was to determine if the change in absolute headache days from baseline to week 24 differed between treatment groups. This objective was assessed using linear regression models, with three pairwise comparisons between treatment groups (Amitriptyline vs. Placebo, Topiramate vs. Placebo, and Amitriptyline vs. Topiramate). The models, and corresponding odds ratios, were adjusted for the two stratification variables (age and baseline number of headache days); Test type: Superiority; p = 0.3553, Regression, Linear — Each comparison was tested using a Bonferroni corrected significance level of 0.017 (0.05/3); Mean Difference (Final Values) = -0.72, 98.3% CI 2-sided [-2.59 to 1.15]
Statistical Analysis 2: Comparison: Topiramate vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.4143, Regression, Linear — Each comparison was tested using a Bonferroni corrected significance level of 0.017 (0.05/3); Median Difference (Final Values) = -0.64, 98.3% CI 2-sided [-2.52 to 1.24]
Statistical Analysis 3: Comparison: Topiramate vs Amitriptyline; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.9038, Regression, Linear — Each comparison was tested using a Bonferroni corrected significance level of 0.017 (0.05/3); Median Difference (Final Values) = -0.08, 98.3% CI 2-sided [-1.68 to 1.52]

4. Secondary Outcome: Tolerability, as Indicated by the Number (Percentage) of Participants That Completed the 24-week Treatment Phase
Description: To assess tolerability, the percentage of subjects who complete the entire 24-week treatment period will be estimated in each of the three groups.
Time Frame: 24 weeks
Population: Tolerability was assessed for all participants included in the primary analysis. Of those randomized, 33 were not included in the primary analysis due to early trial closure.
Measure: Count of Participants; unit: Participants
Arm/Group | Topiramate | Placebo | Amitriptyline
Number analyzed (Participants) | 130 | 66 | 132
Participants | 102 | 59 | 106
Statistical Analysis 1: Comparison: Placebo vs Amitriptyline; Tolerability was assessed by calculating the percent of subjects who completed the entire 24 week treatment period and the corresponding 95% confidence intervals for each treatment group. Concerns regarding tolerability would be raised if the upper bound of a confidence interval was less than 65% or if the percent of subjects who completed the entire 24 week treatment period in either of the active treatment groups was significantly less than the placebo group; Test type: Superiority; p = 0.1557, Fisher Exact; Odds Ratio (OR) = 2.07, 95% CI 2-sided [0.85 to 5.05]
Statistical Analysis 2: Comparison: Topiramate vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0754, Fisher Exact; Odds Ratio (OR) = 2.31, 95% CI 2-sided [0.95 to 5.62]
Statistical Analysis 3: Comparison: Topiramate vs Amitriptyline; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.7611, Fisher Exact; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.49 to 1.62]

5. Secondary Outcome: Occurrence of Treatment Emergent Serious Adverse Events
Description: To determine if amitriptyline or topiramate differ from placebo on the occurrence of treatment emergent serious adverse events.
Time Frame: 24 weeks of the trial
Measure: Number; unit: serious adverse events
Arm/Group | Topiramate | Placebo | Amitriptyline
Number analyzed (Participants) | 145 | 72 | 144
serious adverse events | 4 | 2 | 6
Statistical Analysis 1: Comparison: Placebo vs Amitriptyline; The occurrence of treatment-related SAE's was assessed in two ways: 1) percentage of subjects who experience any treatment-related SAE in each of the three groups was compared using Fishers exact test; 2) rates of treatment-emergent SAS's across the three groups were compared using a Poisson regression model. However, due to the small number of SAEs that were deemed treatment-emergent (4 in AMI, 1 in TPM, 0 in PBO), the parameter estimates did not converge for the Poisson regression model; Test type: Superiority; p = 0.3038, Fisher Exact
Statistical Analysis 2: Comparison: Topiramate vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 3: Comparison: Topiramate vs Amitriptyline; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.2139, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events were collected after the ingestion of at least one dose of study drug through study completion, an average of 24 weeks.
Arm/Group | Topiramate | Placebo | Amitriptyline
Serious Adverse Events (participants affected / at risk) | 4/145 | 2/72 | 6/144
Other Adverse Events (participants affected / at risk) | 111/145 | 51/72 | 106/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate (N=145) | Placebo (N=72) | Amitriptyline (N=144)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic Liver Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate (N=145) | Placebo (N=72) | Amitriptyline (N=144)
Asphasia (Nervous system disorders) | 23 (25) | 7 (9) | 13 (16)
Cognitive Disorder (Nervous system disorders) | 23 (25) | 8 (8) | 14 (18)
Dizziness (Nervous system disorders) | 9 (9) | 1 (2) | 3 (3)
Memory Impairment (Nervous system disorders) | 24 (29) | 7 (8) | 11 (11)
Paresthesia (Nervous system disorders) | 45 (67) | 6 (6) | 10 (10)
Fatigue (General disorders) | 36 (40) | 10 (12) | 43 (48)
Dry Mouth (Gastrointestinal disorders) | 26 (30) | 9 (9) | 36 (45)
Streptococcal Pharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 7 (7)
Upper Respiratory Tract Infection (Infections and infestations) | 18 (19) | 10 (10) | 14 (16)
Mood Altered (Psychiatric disorders) | 14 (16) | 4 (4) | 8 (8)
Decreased Weight (Investigations) | 11 (11) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No